CLINICAL TRIAL: NCT06157125
Title: Assessment of the Association Between Metabolic Associated Fatty Liver Disease MFLD and Glomerulonephritis
Brief Title: Assessment of the Association Between Metabolic Associated Fatty Liver Disease (MFLD) and Biopsy Proved Cases of GN
Acronym: MFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Abd Elkader Anwar, Randa Abd Elkader Anwar, Assiut University
Other Study IDs: MFLD and GN
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Assessment of Patients With Biopsy Proven Primary Glomerulonephritis Above 18 Years of Age for MFLD Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fatty liver disease is a global health concern with a prevalence of about 25% amongst United States. Its increased prevalence is attributed to increase in patients with obesity and metabolic syndrome (1). Diabetes mellitus (DM),obesity, hyperinsulinemia are predisposing factors for fatty liver disease(2). Glomerulonephritis (GN), a complex syndrome encompassing a variety of individual disorders, is associated with significant morbidity and mortality(3). Given its association with hyperlipidaemia, metabolic syndrome and long-term use of steroid there is concern that patients with GN may be at increased risk of fatty liver disease Patients with NS are frequently found to have fatty liver disease even when adjusting for common risk factors(1). It is known that obesity is an independent risk factor for CKD and it is associated with the development of proteinuria and pathologic findings of podocyte hypertrophy and focal segmental glomerular sclerosis even in the absence of diabetes and hypertension . In addition, studies have shown that obesity as well as metabolic syndrome is a strong predictor of the development of fatty liver disease (4) . Hence, clinicians should maintain a high index of suspicion regarding presence of NAFLD in patients with NS

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven primary glomerulonephritis.
* Age >18 years

Exclusion Criteria:

1. Patients with e-GFR<60ml/min/1.73m2
2. Patients with secondary glomerulonephritis
3. Patients with body mass index >35 kg/m2
4. Patients known to be diabetic.
5. Patients known to be hypertensive.
6. Patients with HCV or HBV infection either acute or chronic
7. Patients with acute hepatitis whatever the aetiology
8. Patients with autoimmune diseases

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Patients with biopsy proven primary glomerulonephritis.
  * Age >18 years
  Exclusion Criteria:
  1. Patients with e-GFR<60ml/min/1.73m2
  2. Patients with secondary glomerulonephritis
  3. Patients with body mass index >35 kg/m2
  4. Patients known to be diabetic.
  5. Patients known to be hypertensive.
  6. Patients with HCV or HBV infection either acute or chronic
  7. Patients with acute hepatitis whatever the aetiology
  8. Patients with autoimmune diseases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the association between MFLD and GN | Within 1 year
  Assessment of the association between MFLD and GN

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals nephrology department, Asyut, Egypt

REFERENCES:
- [Background] Amarapurkar D, Kamani P, Patel N, Gupte P, Kumar P, Agal S, Baijal R, Lala S, Chaudhary D, Deshpande A. Prevalence of non-alcoholic fatty liver disease: population based study. Ann Hepatol. 2007 Jul-Sep;6(3):161-3. PMID 17786142
- [Background] Wetmore JB, Guo H, Liu J, Collins AJ, Gilbertson DT. The incidence, prevalence, and outcomes of glomerulonephritis derived from a large retrospective analysis. Kidney Int. 2016 Oct;90(4):853-60. doi: 10.1016/j.kint.2016.04.026. Epub 2016 Jul 15. PMID 27425855
- [Background] Marcuccilli M, Chonchol M. NAFLD and Chronic Kidney Disease. Int J Mol Sci. 2016 Apr 14;17(4):562. doi: 10.3390/ijms17040562. PMID 27089331
- [Result] Onwuzo SS, Hitawala AA, Boustany A, Kumar P, Almomani A, Onwuzo C, Monteiro JM, Asaad I. Prevalence of non-alcoholic fatty liver disease in patients with nephrotic syndrome: A population-based study. World J Hepatol. 2023 Feb 27;15(2):265-273. doi: 10.4254/wjh.v15.i2.265. PMID 36926242